CLINICAL TRIAL: NCT00519441
Title: Gastroesophageal Reflux in Patients With Achalasia
Brief Title: Do Patients Who Have Had Surgery for Achalasia Suffer From Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Luberice (Other)
Responsible Party: Sponsor-Investigator, Kenneth Luberice, Clinical Research Coordinator, University of South Florida
Organization: University of South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 104802
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Reflux
Keywords: laparoscopic Heller myotomy, achalasia, reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Achalasia | interventions — tetrachloroisophthalonitrile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): All patients in the study will have pH studies done in order to determine the degree of reflux after laparoscopic Heller myotomies.
  Interventions: Other: pH study

INTERVENTIONS:
Other: pH study — All patients will have 48 hour pH study
  Other Names: Bravo

SUMMARY:
Patients who have had laparoscopic surgery for the treatment of achalasia will be asked to have pH studies done in order to determine is these patients suffer from reflux after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine if patients who have laparoscopic Heller myotomies for the treatment of achalasia suffer from reflux after the surgery. Patients at our institution who have had surgery for achalasia will be asked to have pH studies done to determine whether or not these patients have reflux.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had laparoscopic Heller myotomies for the treatment of achalasia

Exclusion Criteria:

* Patients under the age of 18 will not be included
* Patients who are receiving anti-reflux therapy will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to determine the degree of post-operative reflux in patients who have had laparoscopic Heller myotomies for the treatment of achalasia. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Cowgill, MD, Principal Investigator — University of South Florida
Locations (1):
- Harbourside Medical Tower, Tampa, Florida, United States